CLINICAL TRIAL: NCT02958670
Title: Imaging Tau Deposition in the Brain of Elderly Subjects
Acronym: Add-Tau
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Collaborators: Avid Radiopharmaceuticals (Industry); Swiss Federal Institute of Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KEK-ZH_Nr_2016-01079_V10.0
Record Dates: First submitted 2016-11-01; First posted 2016-11-08 (Estimated); Last update posted 2023-11-09 (Actual); Status verified 2023-11

CONDITIONS: Mild Cognitive Impairment; Healthy; Alzheimer Disease; Neurocognitive Disorders
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Neurocognitive Disorders | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 18F-AV-1451-PET (Experimental): All subjects receive a Scan for assessment of TAU with the radiotracer 18-F-AV-1451
  Interventions: Other: 18F-AV-1451 (Tau-PET tracer)

INTERVENTIONS:
Other: 18F-AV-1451 (Tau-PET tracer) — Single i.v. administration of 18F-AV-1451 (Tau-PET tracer) and consecutive Positron-Emission-Tomography-Scan

SUMMARY:
Cerebral accumulation of tau and beta-amyloid are major factors of Alzheimer's disease pathology. A novel Positron Emission Tomography (PET) tracer (18-F-AV-1451) now offers the ability to study tau protein deposition in vivo in subjects, in which information on cerebral amyloid deposition has already been gathered. This enables to study effects of tau deposition on neuronal integrity, their relation to effects of beta-amyloid deposition and how this contributes to cognitive impairment or well-being in the elderly.

DETAILED DESCRIPTION:
This is a single-center exploratory observational clinical study combining cross sectional and longitudinal aspects. It contains 18F-AV-1451-PET as an intervention. The primary objective is to measure tau deposition with 18-F-AV1451-PET based on voxel wise or volume based quantitative assessments and to study the effects of Tau deposition on the organism by identification of factors correlating to the measured tau deposition. Study participants will be followed for up to 8 years.

To date cerebral tau pathology in vivo was only estimated by cerebrospinal fluid (CSF) tau or CSF phospho-tau which precludes a study of topical distribution and interplay with Abeta pathology. 18F-AV-1451 offers the chance to visualize tau pathology and to study effects of tau on brain structure, brain physiology and cognitive function. Ideally, these effects are studied in well characterized individuals in whom other important pathological factors are already known.

We therefore plan to study tau pathology measured by 18F-AV-1451 in subjects with already existing data on cerebral amyloid deposition (11C-Pittsburgh Compound C, Flutemetamol). We will be able to relate tau pathology to past and prospective cognitive performance assessed by a detailed neuro¬psychological examination, and we will be able to investigate whether cerebral tau pathology is reflected by peripheral blood biomarkers. For this purpose we will include elderly subjects with various degrees of cognitive performance (cognitively healthy, mild cognitive impairment, dementia) and various degrees of cerebral amyloid deposition (dichotomized or quantitative). We will also include Frontotemporal Lobar Degeneration (FTLD) cases to study tau effects in neurodegenerative disease in the absence of beta-amyloid.

Our hypotheses are the following:

1. We assume that it is possible to identify tau deposition in subjects with and without cerebral Abeta deposition.
2. We hypothesize that tau-deposition will be associated with structural and physiological brain changes and that there are synergistic effects of the amount of tau and Abeta pathology on certain brain regions and on cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Subject belongs to one of the following groups:

   * No cognitive impairment
   * Mild cognitive impairment according to Winblad et al., 2004
   * Clinical diagnosis of dementia due to Alzheimer's disease compatible with DSM IV criteria or revised NINCDS-ADRDA criteria
   * Evidence of neurodegenerative disease other than AD
2. Written informed consent approved by the regulatory authorities
3. Age ≥ 50 years, women must be without childbearing potential
4. Pre-existing PET information (11C-Pittsburgh Compound B, 18F-Flutemetamol) on cerebral amyloid deposition
5. German speaking or sufficient knowledge of German language to perform study assessments
6. Subject is willing and able to name an informant who can give adequate information on the scales where informant input is required

Exclusion Criteria:

1. Evidence for cognitive impairment mainly attributed to a non-neurodegenerative underlying medical condition (e.g. medication, brain tumor, severe heart insufficiency, hepatic encephalopathy)
2. Evidence of larger cerebral infarcts, or lacunes in critical memory structures
3. Disease or other condition with a potential to interfere with study participation
4. Ongoing infection with human immunodeficiency virus (HIV) or any hepatitis virus
5. Active, acute or chronic leukemia
6. Severe illness likely to cause disability that interferes with study procedures in the following years
7. Evidence of acute psychiatric disease (upon clinical decision) which may be a cause of cognitive impairment. Patients with a history of major depression under stable medication may be included. Patients with low dose intake of benzodiazepines may also be included upon clinician's decision
8. Previous or current participation in anti-beta-amyloid or anti-tau therapeutic trials
9. MR exclusion criteria
10. PET exclusion criteria
11. Contraindications against venous puncture
12. Other condition that might pose a risk to the study subject in the opinion of the investigator
13. Exclusion criteria for subproject CSF sampling

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 141 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Volume of Interest (VOI) or Voxel based assessment of 18F-AV-1451-PET-signal | Baseline measurement

OTHER OUTCOMES:
Transition from one clinical state to another (e.g. MCI to AD) worsening of clinical function measured as an increase in CDRSOB-score of one | up to two years
Neuropsycholgical test performance | up to two years
Magnetresonance Tomography (MR) readouts | Baseline and two years
Blood and CSF-biomarker-read outs | Baseline and two years

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Hock, Prof.Dr. med, Principal Investigator — Professor for Biological Psychiatry, Institute for Regenerative Medicine, University of Zurich
Locations (1):
- Institute for Regenerative Medicine (IREM), Schlieren, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No